CLINICAL TRIAL: NCT05497895
Title: A Randomized Controlled Clinical Trial for the Assessment of Clinical Efficacy of Topical Application of 5% Thymoquinone Gel for Gingivitis Patients
Brief Title: The Assessment of Clinical Efficacy of Topical Application of 5% Thymoquinone Gel for Gingivitis Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ahmad Almehmadi, Associate Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAAU
Record Dates: First submitted 2022-06-17; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Gingivitis
Keywords: Gingivitis; THYMOQUINONE; Clinical Trial
MeSH Terms: conditions — Gingivitis | interventions — thymoquinone; Gels

STUDY DESIGN:
Intervention Model Description: DESIGN: Double-blinded, parallel, randomized controlled clinical trial. SETTING: Faculty of Dentistry, King Abdulaziz University, and Qassim University, Saudi Arabia PARTICIPANTS AND METHODS: This trial will enroll 63 participants with age group between 18-40 years attending the outpatient clinics of Faculty of dentistry, Qassim University, Saudi Arabia with confirmed clinical diagnosis of gingivitis. The enrolled subjects will be categorized in three groups: Group I-TQ gel with SRP, Group II-Placebo with SRP, and Group III-SRP alone and clinical outcomes will be measured at baseline and two-week follow-up visit.
  MAIN OUTCOME MEASURES: Plaque Index (PI), Papillary Bleeding Index (PBI) and any adverse events with TQ gel categorized as mild, moderate, and severe.
  SAMPLE SIZE: 63 patients. Group I (n=21); Group II (n=21); Group III (n=21)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (SRP and TQ gel) (Experimental): In Group I patients, the lipid based TQ gel (5%) will be applied topically to the affected areas, twice daily for two weeks following SRP. The investigator performs the treatment of gingivitis based on the patient's response to therapy. For home care, the patients will be instructed to clean and dry the affected area prior to the gel application and hands will be washed prior and after its application. The patients will be instructed to not eat for 30 minutes following its application
  Interventions: Biological: 5% thymoquinone (TQ) gel
- Group II (SRP and Placebo) (Placebo Comparator): In Group II patients, the placebo gel will be applied topically to the affected areas, twice daily for two weeks following SRP. The investigator performs the treatment of gingivitis based on the patient's response to therapy. For home care, the patients will be instructed to clean and dry the affected area prior to the gel application and hands will be washed prior to and after its application. The patients will be instructed to not eat for 30 minutes following its application
  Interventions: Biological: SRP and placebo
- Group III (Only SRP and one stage prophylaxis) (Active Comparator): The Group III patients will be subjected to one-stage oral prophylaxis.
  Interventions: Procedure: Only SRP-one stage prophylaxis

INTERVENTIONS:
Biological: 5% thymoquinone (TQ) gel — Mode of Administration In Group I patients, the lipid based TQ gel (5%) will be applied topically to the affected areas, twice daily for two weeks following SRP. The investigator performing the treatment of gingivitis based on the patient's response to therapy. For home care, the patients will be instructed to clean and dry the affected area prior to the gel application and hands will be washed prior and after its application. The patients will be instructed to not eat for 30 minutes following its application.
  Arms: Group I (SRP and TQ gel)
Biological: SRP and placebo — In Group II patients, the placebo gel will be applied topically to the affected areas, twice daily for two weeks following SRP. The investigator performs the treatment of gingivitis based on the patient's response to therapy. For home care, the patients will be instructed to clean and dry the affected area prior to the gel application and hands will be washed prior to and after its application. The patients will be instructed to not eat for 30 minutes following its application
  Arms: Group II (SRP and Placebo)
Procedure: Only SRP-one stage prophylaxis — The Group III patients will be subjected to one-stage oral prophylaxis.
  Arms: Group III (Only SRP and one stage prophylaxis)

SUMMARY:
Gingival diseases occur commonly in the global population and herbal products for its intervention have limited body of research evidence. This study to evaluate the clinical efficacy of 5% thymoquinone (TQ) gel as an adjunct to scaling and root planing (SRP) in patients diagnosed with gingivitis.

OBJECTIVE: To evaluate the efficacy of 5% TQ gel using a novel liposome drug delivery as a topical application following SRP in gingivitis patients.

DESIGN: Double-blinded, parallel, randomized controlled clinical trial. SETTING: Faculty of Dentistry, King Abdulaziz University, and Qassim University, Saudi Arabia

DETAILED DESCRIPTION:
This randomized controlled clinical trial will be conducted to evaluate of clinical efficacy of TQ gel (5%) as an adjunct to SRP in patients with gingivitis (n=63). The patients will be recruited from the Faculty of Dentistry, Qassim University and the subjects will be divided into three groups and include Group I (SRP+TQ gel), Group II (SRP+Placebo), and Group III (Only SRP-one stage prophylaxis). The subjects will be given an explanation of the purpose of the study; informed consent will be obtained in a written format. This clinical trial will be performed in accordance with the ICH (International Conference on Harmonization-E6 'Guideline for Good Clinical Practice') and Helsinki Declaration 1975, as revised in 2000. The study protocol was approved by the Institutional Review Board, Qassim University, Saudi Arabia (IRB No: EAC 104-2018). The complete oral diagnosis will be performed during the screening visit by clinical assessment and periapical radiographs may be indicated to obtain a definitive diagnosis, The periodontal charting will be performed and recorded in the patient's case record. The participants will be consecutively enrolled with the following inclusion and exclusion criteria.

Preparation of Lipid-based TQ gel formulation (5%):

Thymoquinone extract (Sigma Aldrich extract-Product No:03416) was obtained in crystalline form.

Mode of Administration In Group I patients, the lipid-based TQ gel (5%) will be applied topically to the affected areas, twice daily for two weeks following SRP. The investigator will perform the treatment of gingivitis based on the patient's response to therapy. For home care, the patients will be instructed to clean and dry the affected area prior to the gel application and hands to be washed prior to and after its application. The patients would be instructed to not eat for 30 minutes following its application. The same will be done for Group II patients who were treated with SRP followed by a placebo gel application in the affected areas. The Group III patients will be subjected to one-stage oral prophylaxis. It will be a double-blinded clinical trial as the patients would not be made aware of which gel preparation was given to them and the principal investigators would not be aware of the patient's group while performing clinical measurements, whereas the operator performed SRP and gel application.

Treatment Compliance A diary card will be given to all the patients along with instructions on filling the card and reminders to bring it on subsequent visits will be mentioned. The principal investigator will ensure that each patient used at least 75% and not more than 125% of the study drug over the course of the study period. The drug accountability i.e., receipt, dispensing, and return of the drug) will be performed either by the principal investigator or his designee. The assessment of the primary endpoint will be based on the clinical scoring conducted on a weekly basis till the end of the study.

Clinical Evaluation The clinical parameters such as plaque index (PI) and papillary bleeding index (PBI) will be evaluated for all the patients at the appropriate follow-up intervals. The parameters will be evaluated by two independent examiners. The adverse events, if any with the administration of TQ gel will be monitored and it would be graded as per the intensity as mild, moderate, and severe.

Discontinuation of Treatment In case of adverse events with the use of the study drug, the patients would be withdrawn from therapy or clinical assessment. Also, when the patients suffer from significant illness or undergo surgery during the course of the study, they would be withdrawn from the trial. The non-compliant patients who did not adhere to the study protocol or for other justifiable reasons were withdrawn from the current clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* • Patient diagnosed with gingivitis (Probing<3mm with bleeding on probing ≥10% of sites) (Trombelli, Farina et al. 2018)

  * Minimum twenty teeth in the oral cavity
  * Age: 18-40 years

Exclusion Criteria:

* • Patients with systemic diseases that have an association with periodontal diseases like diabetes, cardiovascular diseases, blood dyscrasias, or diseases of immune system and would require antibiotics prior to dental treatment

  * Patients who received antibiotic therapy in the last 3 months prior to the trial
  * Pregnant or lactating females
  * Patients treated with drugs such as antacids, warfarin or cyclosporine
  * Presence of overhanging restorations or other contributing factors to periodontal disease
  * Allergy to Nigella sativa and/or TQ

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Plaque index | 2 weeks
  The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth:
  0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Papillary bleeding index | 2 weeks
  This index permits both immediate evaluation of the patient's gingival condition and his motivation, based upon the actual bleeding tendency of the gingival papillae. A periodontal probe is inserted into the gingival sulcus at the base of the papilla on the mesial aspect, and then moved coronally to the papilla tip. This is repeated on the distal aspect of the papilla. The intensity of any bleeding is recorded as: Score 0 - no bleeding; Score 1 - A single discreet bleeding point; Score 2 - Several isolated bleeding points or a single line of blood appears; Score 3 - The interdental triangle fills with blood shortly after probing; Score 4 - Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.

SECONDARY OUTCOMES:
Number of participants with drug related adverse events | Duration of the clinical trial
  Reported during the trial and on clinical assessment
Number of participants non compliant/withdraw from the study | Duration of the clinical trial
  Reported during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad AlMehmadi, Principal Investigator — King Abdul Aziz University
Locations (1):
- Qassim University, Buraidah, Saudi Arabia

REFERENCES:
- [Background] Abou Sulaiman AE, Shehadeh RMH. Assessment of Total Antioxidant Capacity and the Use of Vitamin C in the Treatment of Non-Smokers With Chronic Periodontitis. J Periodontol. 2010 Nov;81(11):1547-54. Adair JG. The Hawthorne effect: A reconsideration of the methodological artifact. J Appl Psychol. 1984;69(2):334-45. Akalin FA, Toklu E, Renda N. Analysis of superoxide dismutase activity levels in gingiva and gingival crevicular fluid in patients with chronic periodontitis and periodontally healthy controls. J Clin Periodontol. 2005 Mar;32(3):238-43. Albandar JM, Brown LJ, Brunelle JA, Löe H. Gingival State and Dental Calculus in Early-Onset Periodontitis. J Periodontol. 1996 Oct;67(10):953-9. Al-Bayaty FH, Kamaruddin AA, Ismail MohdA, Abdulla MA. Formulation and Evaluation of a New Biodegradable Periodontal Chip Containing Thymoquinone in a Chitosan Base for the Management of Chronic Periodontitis. J Nanomater. 2013;2013:1-5. Al Wafi H. Benefits of Thymoquinone, a Nigella SativaExtract in Preventing Dental Caries Initiation and Improving Gingival Health. ProQuest LLC [Internet]. 2014; Available from: search.proquest.com Chapple ILC, Brock GR, Milward MR, Ling N, Matthews JB. Compromised GCF total antioxidant capacity in periodontitis: cause or effect? J Clin Periodontol [Internet]. 2007 Feb [cited 2020 Mar 26];34(2). Available from: http://doi.wiley.com/10.1111/j.1600-051X.2006.01029.x D'Aiuto F, Nibali L, Parkar M, Patel K, Suvan J, Donos N. Oxidative stress, systemic inflammation, and severe periodontitis. J Dent Res. 2010 Nov;89(11):1241-6. Feil PH, Grauer JS, Gadbury-Amyot CC, Kula K, McCunniff MD. Intentional use of the Hawthorne effect to improve oral hygiene compliance in orthodontic patients. Journal of dental education. 2002 Oct 1;66(10):1129-35. Idrees MM, Azzeghaiby SN, Hammad MM, Kujan OB. Prevalence and severity of plaque-induced gingivitis in a Saudi adult population. Saudi Med J. 2014 Nov;35(11):1373-7. Kataoka K, Ekuni D, Tomofuji T, Irie K, Kunitomo M, Uchida Y, et al. Visualization of Oxidative Stress Induced by Experimental Periodontitis in Keap1-Dependent Oxidative Stress Detector-Luciferase Mice. Int J Mol Sci. 2016 Nov 16;17(11):1907. Kandwal A, Mamgain R, Mamgain P. Comparative evaluation of turmeric gel with 2% chlorhexidine gluconate gel for treatment of plaque induced gingivitis: A randomized controlled clinical trial. AYU Int Q J Res Ayurveda. 2015;36(2):145. Kapil H, Suresh DK, Bathla SC, Arora KS. Assessment of clinical efficacy of locally delivered 0.2% Thymoquinone gel in the treatment of periodontitis. Saudi Dent J. 2018 Oct;30(4):348-54. Król K. [Reactive oxygen species and antioxidant mechanisms in the pathogenesis of periodontitis]. Ann Acad Med Stetin. 2004;50(2):135-48. Löe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov;38(6):610-6. Mariod AA, Ibrahim RM, Ismail M, Ismail N. Antioxidant activity and phenolic content of phenolic rich fractions obtained from black cumin (Nigella sativa) seedcake. Food Chem. 2009 Sep;116(1):306-12. Ozdemir H, Kara MI, Erciyas K, Ozer H, Ay S. Preventive effects of thymoquinone in a rat periodontitis model: a morphometric and histopathological study: Effects of thymoquinone in a rat periodontitis model. J Periodontal Res. 2012 Feb;47(1):74-80. Pihlstrom BL. Periodontal risk assessment, diagnosis and treatment planning. Periodontol 2000. 2001;25:37-58. Pradeep AR, Rao NS, Bajaj P, Agarwal E. 8-Isoprostane: A lipid peroxidation product in gingival crevicular fluid in healthy, gingivitis and chronic periodontitis subjects. Arch Oral Biol. 2013 May;58(5):500-4. Ragheb A, Attia A, Eldin W, Eibarbry F, Gazarin S, Shoker A. The protective effect of thymoquinone, an anti-oxidant and anti-inflammatory agent, against renal injury: a review. 2009;20(5):741. Saxer UP, Mühlemann HR. [Motivation and education]. Schweiz Monatsschrift Zahnheilkd Rev Mens Suisse Odonto-Stomatol. 1975 Sep;85(9):905-19. Sercombe L, Veerati T, Moheimani F, Wu SY, Sood AK, Hua S. Advances and Challenges of Liposome Assisted Drug Delivery. Front Pharmacol [Internet]. 2015 Dec 1 [cited 2020 Mar 26];6. Available from: http://journal.frontiersin.org/article/10.3389/fphar.2015.00286 Trombelli L, Farina R, Silva CO, Tatakis DN. Plaque-induced gingivitis: Case definition and diagnostic considerations. J Periodontol. 2018 Jun;89:S46-73.